CLINICAL TRIAL: NCT01034020
Title: Effects of Nicotine on Elements of Attentions in Smokers and Nonsmokers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Purpose: Treatment
Other Study IDs: 999906409; 06-DA-N409
Record Dates: First submitted 2009-12-16; First posted 2009-12-17 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2010-09-22

CONDITIONS: Substance Related Disorder; Nicotine Dependence
Keywords: Nasal Spray; Attention Network Test; Continuous Performance Test; Attentional Blink Test
MeSH Terms: conditions — Substance-Related Disorders; Tobacco Use Disorder | interventions — Nicotine

INTERVENTIONS:
Drug: Nicotine

SUMMARY:
Background:

- Many cigarette smokers claim that smoking helps them stay alert and improves their concentration, and have reported problems in attention and concentration after quitting smoking. Some research has indicated that nicotine can enhance certain aspects of attention and memory in humans. However, more research is needed to determine how nicotine affects different elements of the brain's ability to pay attention. Knowing which aspects of attention are affected by nicotine may help produce new medications and therapies to help people successfully stop smoking.

Objectives:

* To investigate the dose-related effects of nicotine on the ability to pay attention in smokers and nonsmokers.
* To compare the effects of nicotine in smokers and nonsmokers.

Eligibility:

- Individuals between 18 and 50 years of age who are either current smokers (at least 15 cigarettes per day on average for at least 2 years) or healthy, nonsmoking volunteers.

Design:

* The study will consist of one training session and three testing sessions. Each session will last about 2 hours.
* The training session will introduce participants to the study tests and evaluate their tolerance of the two levels of nicotine nasal spray used in the study. Smokers will receive the higher dose of nicotine to introduce them to the effects of the spray. Nonsmokers will be given first the lower dose of the spray, followed by higher dose at least 30 minutes later. Nonsmoking participants who cannot tolerate the higher dose will not continue in the study.
* At the start of each testing session, smokers will have one cigarette to standardize the time of the most recent exposure to nicotine.
* During the testing sessions, participants will receive a placebo spray, a lower dose of nicotine, or a higher dose of nicotine, and then will be asked to perform tests that evaluate mood, attention, and performance.

DETAILED DESCRIPTION:
Objective: The primary objective of this study is to investigate the dose-related effects of nicotine on various elements of attention in smokers and nonsmokers. Because no published study, to our knowledge, has reported the effects of nicotine on the ANT and ABT, we will include the CPT, a task shown to be sensitive to nicotine, as a positive control. A secondary aim is to compare the subjective and physiological effects of nicotine between smokers and nonsmokers.

Study Population: 50 smokers for a total of 30 completers (15 women, 15 men) and up to 50 nonsmokers for a total of 30 completers (15 women, 15 men).

Design: Placebo-controlled, between-groups comparison of smokers and nonsmokers. Participants will attend three experiemental sessions; a single dose of nicotine nasal spray (0, 0.5, or 1.5 mg) will be administered at each session.

Outcome Measures: Primary outcome measures will be accuracy and/or response time on the three attention tests, ANT, CPT, and ABT. Secondary outcome measures include responses to the PANAS, VAS items, and vital signs (heart rate and blood pressure). Participant demographics and smoking history will be reported using descriptive statistics.

ELIGIBILITY:
* INCLUSION CRITERIA: Smokers

  1. be men and women 18-50 years old
  2. report smoking at least 15 cigarettes per day on average for at least 2 years
  3. have a urine cotinine level greater than or equl to 200 ng/ml
  4. have an estimated IQ score greater than or equal to 85
  5. be medically and psychologically healthy as determined by screening criteria

     EXCLUSION CRITERIA: Smokers

  <!-- -->

  1. be interested in reducing or quitting tobacco use
  2. have been treated for nicotine dependence in the past 3 months 3) report a history of drug or alcohol dependence

  4) report consumption of more than 15 alcoholic drinks per week during the past month

  5) report use of marijuana more than once per week during the past month

  6) report use of any illicit drug, other than marijuana, during the past 6 months

  7) be currently using any medication that would interfere with the protocol

  8) be under the influence of a drug or alcohol at experimental sessions

  9) be pregnant or nursing

  10) be HIV positive.

INCLUSION CRITERIA: Nonsmokers

1. be men and women 18-50 years old
2. report smoking less than 10 cigarettes in their life
3. have a urine cotinine level less than 30 ng/ml
4. have an estimated IQ score greater than or equal to 85
5. be medically and psychologically healthy as determined by screening criteria

EXCLUSION CRITERIA: Nonsmokers

1. report use of any tobacco products in the past 3 years
2. report a history of drug or alcohol dependence
3. report consumption of more than 15 alcoholic drinks per week during the past month
4. report use of marijuana more than once per week during the past month
5. report use of any illicit drug, other than marijuana, during the past 6 months
6. be currently using any medication that would interfere with the protocol
7. be under the influence of a drug or alcohol at experimental sessions
8. be pregnant or nursing
9. be HIV positive.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Estimated)
Dates: Start 2006-02-14; Primary Completion 2009-11-03 (Actual); Study Completion 2009-11-03 (Actual)

PRIMARY OUTCOMES:
Pharmacodynamics, changes in cognitive function

SECONDARY OUTCOMES:
Changes in subjective mood, changes in cardiovascular measures

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute on Drug Abuse, Biomedical Research Center (BRC), Baltimore, Maryland, United States

REFERENCES:
- [Background] Bancroft A, Levin ED. Ventral hippocampal alpha4beta2 nicotinic receptors and chronic nicotine effects on memory. Neuropharmacology. 2000 Oct;39(13):2770-8. doi: 10.1016/s0028-3908(00)00099-x. PMID 11044746
- [Background] Benowitz NL, Jacob P 3rd. Nicotine and cotinine elimination pharmacokinetics in smokers and nonsmokers. Clin Pharmacol Ther. 1993 Mar;53(3):316-23. doi: 10.1038/clpt.1993.27. PMID 8453850
- [Background] Bizarro L, Patel S, Murtagh C, Stolerman IP. Differential effects of psychomotor stimulants on attentional performance in rats: nicotine, amphetamine, caffeine and methylphenidate. Behav Pharmacol. 2004 May;15(3):195-206. PMID 15187577